CLINICAL TRIAL: NCT01559493
Title: Comparison of Fractional Flow Reserve Versus Instant Wave-Free Ratio for Assessment of Coronary Artery Stenosis Severity in Routine Practice
Brief Title: Fractional Flow Reserve (FFR) Versus Instant Wave-Free Ratio (iFR)
Status: Completed | Type: Observational
Sponsor: NHS National Waiting Times Centre Board (Other)
Collaborators: Golden Jubilee National Hospital (Other Government); Catharina Ziekenhuis Eindhoven (Other); Onze Lieve Vrouw Hospital (Other); Stockholm South General Hospital (Other); Brno University Hospital (Other); Stanford University (Other)
Responsible Party: Principal Investigator, Prof. Keith G. Oldroyd, Consultant Cardiologist, NHS National Waiting Times Centre Board
Other Study IDs: Version F 2nd Jan 2012
Record Dates: First submitted 2012-02-14; First posted 2012-03-21 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Coronary Artery Disease; Plaque, Atherosclerotic
Keywords: atherosclerotic lesion assessment
MeSH Terms: conditions — Coronary Artery Disease; Plaque, Atherosclerotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FFR; iFR: Interventional Cardiology, Pressure wire, fractional flow reserve, coronary flow measurement

SUMMARY:
Comparison of Fractional Flow Reserve versus instant Wave-Free Ratio for assessment of coronary artery stenosis severity in routine practice

* To compare FFR to iFR in arbitrary consecutive patients referred for percutaneous coronary intervention (PCI).
* To investigate the influence of hyperemia on iFR.
* To test reproducibility of iFR and FFR.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients undergoing FFR assessment for standard clinical indications.

Exclusion Criteria:

* prior CABG
* extremely tortuous, calcified lesions
* coronary artery occlusion
* acute MI within 5 days

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The aim of the present study is to strengthen the results of retrospective comparisons of iFR with FFR by conducting a prospective study in 200 consecutive, unselected patients from 5 different centers.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Comparison of Fractional Flow Reserve vs. instant Wave-Free Ratio for assessment of coronary artery stenosis severity in routine practice | 30 days
  In this prospective, multicenter, international investigation, all consecutive patients in 5 centers, referred for PCI will be included. FFR will be submitted for one vessel in each patient - this will be the first vessel in which the FFR is performed. Measurements will be performed in duplicate. iFR will be calculated for all lesions for which an FFR measurement is submitted. In addition, iFR and FFR will be compared retrospectively in 1000 patients who had FFR measurements in the recent past

SECONDARY OUTCOMES:
iFR at rest vs iFr during hyperemia | 30 days
  iFR is said to be independent of hyperemia. Accordingly a secondary outcome of this study will be a paired comparison of iFR at rest vs iFr with adenosine induced hyperemia.
Repeatability of iFr and FFR | 30 days
  To test repeatability of iFR and FFR

CONTACTS AND LOCATIONS:
Overall Officials: Prof Keith G. Oldroyd, Principal Investigator — Golden Jubilee National Hospital; Prof Colin Berry, MD, Principal Investigator — Golden Jubilee National Hospital
Locations (5):
- Stanford University, Stanford, California, United States
- Cardiovascular Center Aalst, Aalst, Belgium
- University Hospital Brno, Brno, Czechia
- Catharina Ziekenhuis, Eindhoven, Netherlands
- Stockholm South Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Berry C, van 't Veer M, Witt N, Kala P, Bocek O, Pyxaras SA, McClure JD, Fearon WF, Barbato E, Tonino PA, De Bruyne B, Pijls NH, Oldroyd KG. VERIFY (VERification of Instantaneous Wave-Free Ratio and Fractional Flow Reserve for the Assessment of Coronary Artery Stenosis Severity in EverydaY Practice): a multicenter study in consecutive patients. J Am Coll Cardiol. 2013 Apr 2;61(13):1421-7. doi: 10.1016/j.jacc.2012.09.065. Epub 2013 Feb 6. PMID 23395076